CLINICAL TRIAL: NCT00399412
Title: Further Research on Human Feasibility of a Subcutaneous Implantable Defibrillator (S-ICD)- ECG Signal Collections From Various Patient Groups Whilst Attending Outpatient Follow-up
Brief Title: ECG Signal Collection From Long QT Syndrome, Wide QRS Complexes, Heart Failure, and Cardiac Resynchronization Patients
Status: Completed | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: DN-05291
Record Dates: First submitted 2006-11-10; First posted 2006-11-14 (Estimated); Last update posted 2017-02-16 (Actual); Status verified 2009-10

CONDITIONS: Long QT Syndrome; Wide QRS Complexes; Heart Failure; Cardiac Resynchronisation
Keywords: S-ICD; ICD; ECG signals; Resting
MeSH Terms: conditions — Long QT Syndrome; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- LQTS: Long QT syndrome
  Interventions: Device: subcutaneous ICD
- HF: Heart Failure
  Interventions: Device: subcutaneous ICD
- CRT: Cardiac Resynchronization Therapy
  Interventions: Device: subcutaneous ICD
- Wide QRS: QRS > 120 milliseconds
  Interventions: Device: subcutaneous ICD

INTERVENTIONS:
Device: subcutaneous ICD

SUMMARY:
The purpose of this study is to collect surface electrograms from standard and several non-standard configurations in patients with long QT syndrome, heart failure, cardiac resynchronization therapy or wide QRS during a routine outpatient assessment. The ECGs collected will be used as test signals by the sponsor for the development of a subcutaneous implantable defibrillator

DETAILED DESCRIPTION:
The objective of this study is to record standard ECG signals is each of the 4 patient populations together with signals from 4 non-standard surface positions when these patients attend the outpatient department for follow-up. The non-standard electrode positions mimic the positions of the subcutaneous electrodes of the subcutaneous implantable defibrillator (S-ICD) system in development by Cameron Health.

The collection of these signals will allow bench testing of the algorithms proposed for the S-ICD system. Additionally, it will allow a comparison of the response of different defibrillators to these same signals to asses how each would treat a particular rhythm.

ELIGIBILITY:
Inclusion Criteria:

* Patients attending the outpatient for routine follow-up for their cardiac disease or to have an implanted device follow-up

Exclusion Criteria:

* Patients unable or unwilling to provide informed consent
* Any condition which precludes the subject's ability to comply with the study requirements, including completion of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with long QT syndrome, heart failure, cardiac resynchronization therapy or wide QRS.
Sampling Method: Non-Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2006-11; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew A Grace, MD PhD, Principal Investigator — Papworth Hospital NHS Trust
Locations (1):
- Papworth Hospital NHS Trust, Papworth Everard, Cambridge, United Kingdom